CLINICAL TRIAL: NCT01391351
Title: Search for Predictors of Therapeutic Response in Patients With Carcinoma of the Ovary, the Fallopian Tube or Peritoneal Serous-type Advanced
Brief Title: Search for Predictors of Therapeutic Response in Ovarian Carcinoma
Acronym: miRSa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: miRSa
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Carcinoma of the Ovary; Fallopian Tube Cancer; Peritoneal Serous-type Advanced Stage
Keywords: carcinoma of the ovary, the fallopian tube or peritoneal serous-type advanced stage; chemotherapy with Taxol and Carboplatin; predictors of therapeutic response; serum miRNA; identification of polymorphisms or SNPs (Single Nucleotide Polymorphism)
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taxol and carboplatin (Other): blood samples in patients receiving Taxol and carboplatin chemotherapy
  Interventions: Other: blood samples
- Taxol, carboplatin and avastin (Other): blood samples in patients receiving Taxol, carboplatin chemotherapy with avastin
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — blood samples in patients receiving Taxol and carboplatin chemotherapy :
  * On Day 1 of the first course of chemotherapy
  * On Day 1 of the second course of chemotherapy
  * Before the surgery, if programmed via J1 or the fourth cycle of chemotherapy
  * At the end of chemotherapy
  Arms: Taxol and carboplatin
Other: blood samples — blood samples in patients receiving Taxol and carboplatin chemotherapy with avastin:
  * On Day 1 of the first course of chemotherapy
  * On Day 1 of the second course of chemotherapy
  * Before the surgery, if programmed via J1 or the fourth cycle of chemotherapy
  * At the end of chemotherapy
  Arms: Taxol, carboplatin and avastin

SUMMARY:
In order to search for predictors of response to chemotherapy in patients with ovarian carcinoma of the ovary, the fallopian tube or peritoneal serous-type advanced stage, we will define the comparative profiles of miRNA expression of serum polymorphisms and determine differential in 2 patient populations (with or without recurrence 6 months after completion of chemotherapy) with (i) the miRNA profile of serum before treatment and (ii) identification of polymorphisms or SNP (Single Nucleotide Polymorphism) in particular genes involved in the metabolism of chemotherapy agents In the case of miRNA, expression profiles will also be studied during the first course in response to chemotherapy. Indeed, the miRNA profile of serum may be different at baseline among the 2 types of populations (or non-recurrence at 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer of the ovary, peritoneum or of the fallopian tube
* Stage III or IV
* Cancer of serous histology
* Patients of any chemotherapy naive
* Patients should receive treatment with chemotherapy for first line by Taxol- Carboplatin. Avastin is authorized in concomitant.
* An initial surgery or through authorized
* Patients who signed informed consent
* Patients over the age of 18 years

Exclusion Criteria:

* Patients being treated for another cancer chemotherapy and / or hormone therapy
* Patients receiving other chemotherapy Taxol-carboplatin associated or not to avastin
* Patients under guardianship
* Previous history of pelvic radiotherapy
* History of malignancy blood

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-06; Primary Completion 2015-11 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
search for predictors of response to chemotherapy | 12 months after beginning treatment
  the search for predictors of response to chemotherapy in patients with carcinoma of the ovary, the fallopian tube or peritoneal serous-type advanced by using (i) the miRNA profile of serum before treatment with chemotherapy and (ii) the identification of polymorphisms or SNPs (Single Nucleotide polymorphism) in particular genes involved in the metabolism of chemotherapy agents

SECONDARY OUTCOMES:
profiling miRNA expression | 1 month
  - Characterization of the response to treatment with profiling miRNA expression after the first course of chemotherapy in patients with carcinoma of the ovary, the fallopian tube or peritoneal serous-type advanced
study of changes in serum miRNA expression | 6 months
  - The study of changes in serum miRNA expression identified as predictive of tumor response during chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY-LOBBEDEZ, PD, Principal Investigator — Centre François Baclesse; Sophie KRIEGER, MD, Principal Investigator — Centre François Baclesse
Locations (7):
- France (7):
  - Centre Eugène Marquis, Rennes, Brittany Region
  - Centre François BACLESSE, Caen, Calvados
  - Centre Réné Gauducheau, Nantes, Loire-Atlantique
  - Centre Oscar LAMBRET, Lille, Nord
  - Centre Henri Becquerel, Rouen, Seine Maritime
  - Institut de cancerologie de la loire, Angers
  - Institut CURIE, Paris